CLINICAL TRIAL: NCT06412744
Title: Determination of the Iodine Status in Pregnant Women in the Netherlands. Are Current Iodine Intake Recommendations Still Adequate?
Brief Title: Determination of the Iodine Status in Pregnant Women in the Netherlands.
Acronym: JOZO
Status: Terminated | Type: Observational
Why Stopped: Difficulties finding participants
Sponsor: Maastricht University Medical Center (Other)
Collaborators: National Institute for Public Health and the Environment (RIVM) (Other Government)
Responsible Party: Sponsor
Other Study IDs: NL70677.068.19; NL8297 (Registry Identifier: NL trial register (NTR))
Record Dates: First submitted 2022-12-16; First posted 2024-05-14 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-05

CONDITIONS: Pregnancy Related; Healthy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood (only plasma and serum is stored) Urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Total cohort: No intervention, all participants undergo the same measurements

SUMMARY:
Study to determine iodine status in dutch pregnant women

DETAILED DESCRIPTION:
Rationale: Adequate dietary iodine intake is essential to thyroid hormone synthesis, which is key for normal growth, development and metabolism. During pregnancy, maternal iodine needs are increased (recommended intake: 175 µg/day) and iodine deficiency during pregnancy affects brain and cognitive development of the foetus and might lead to pregnancy complications. Despite the use of iodized salt, it has been shown that iodine intake in the Netherlands is declining. Importantly, a recent small study in Groningen indicated a high prevalence of iodine deficiency during pregnancy (83% of participants) which was not completely restored by 16-week iodine supplementation (150 ug/d). Also in other Western European countries (i.e. Belgium, U.K., North Ireland, Sweden, Denmark and Austria) low median urinary concentrations of iodine (73-124 ug/L) have been observed in pregnant women. Notably, most studies collected spot-urine samples and a 24h urine collection, the golden standard for determination of iodine status, is lacking. Therefore, here it is proposed to measure 24h median urinary iodine concentration corrected for urinary volume and creatinin levels in pregnant women, and compare these values with Thyroglobulin (Tg)-concentrations in serum as measure for iodine intake over a longer period of time. It is hypothesised that the iodine status of pregnant women in The Netherlands is lower than the national recommended intake for this target group.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 18-45y old
* in first 16 weeks of pregnancy
* pregnant of singleton

Exclusion Criteria:

* Thyroid-disease or any other metabolic disease
* kidney disease
* twin-pregnancy

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy pregnant women, under 16 weeks of gestational age living in the Netherlands
Sampling Method: Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2020-10-06 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Median urinary iodine excretion (µg/d) | At baseline measurement
  Median urinary iodine excretion (µg/d)

SECONDARY OUTCOMES:
Thyroglobulin and thyroglobulin antibody concentrations in blood serum | At baseline measurement
  Thyroglobulin and thyroglobulin antibody concentrations in blood serum
Creatinin concentration in urine | At baseline measurement
  Creatinin concentration in urine
Urinary volume | At baseline measurement
  Urinary volume
Smoking status (smoking is interfering with iodine metabolism) | At baseline measurement
  Smoking status (smoking is interfering with iodine metabolism) Yes/no
Vegan/Vegetarian y/n (soy is competitive for iodine on thyroid) | At baseline measurement
  Vegan/Vegetarian y/n (soy is competitive for iodine on thyroid)
Nutritional intake specifically related to iodine intake (questionnaire) | At baseline measurement
  Nutritional intake specifically related to iodine intake (questionnaire) Iodine specific ffq
Intake other relevant micronutrients for pregnant | At baseline measurement
  Intake other relevant micronutrients for pregnant

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht UMC+, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided